CLINICAL TRIAL: NCT00306657
Title: Normal Tension and Chronic Open Angle Glaucoma, Cerebrospinal Fluid Composition in Subarachnoid Space of Affected Optic Nerves
Brief Title: Normal Tension and Chronic Open Angle Glaucoma and Cerebrospinal Fluid Composition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kantonsspital Aarau (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005/057
Record Dates: First submitted 2006-03-23; First posted 2006-03-24 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2007-04

CONDITIONS: Glaucoma Open-Angle
Keywords: Glaucoma Open-Angle; Normal tension glaucoma progressive; chronic open angle glaucoma progressive; optic nerve sheath fenestration; cerebrospinal fluid; Beta-Trace Protein
MeSH Terms: conditions — Glaucoma, Open-Angle

INTERVENTIONS:
Procedure: Optic nerve sheath fenestration

SUMMARY:
Normal tension glaucoma (NTG) and chronic open angle glaucoma (COAG) occurring progressively with optimal conventional or intraocular pressure reducing surgery are still unsolved problems in ophthalmology. The investigators would like to investigate whether or not the composition of cerebrospinal fluid (CSF) surrounding the optic nerve (ON) in these patients is pathologic under certain conditions. They therefore compare the CSF taken during optic nerve sheath fenestration with the CSF taken during a lumbar puncture. The investigators' hypothesis is that, in patients with NTG and COAG, the composition of CSF surrounding the affected ON plays an important role in promoting progressive visual function loss.

DETAILED DESCRIPTION:
We will recruit 30 patients with progressive visual function loss, due to Normal tension glaucoma (NTG) or chronic open angle glaucoma (COAG), despite optimal conventional or intraocular pressure reducing surgery treatment so far. We will proceed with an optic nerve sheath fenestration (ONSF) (according to the studies in the literature, e.g. Wax MB, Barrett DA, Hart WM Jr, Custer PL. Optic nerve sheath decompression for glaucomatous optic neuropathy with normal intraocular pressure. Arch Ophthalmol. 1993;111(9):1219-28.) and compare the cerebrospinal fluid (CSF) taken from the subarachnoid space (SAS) of the optic nerve (ON) with the CSF taken during a lumbar puncture, on the same day. Concentrations of neurobioactive substances will especially be studied. Visual acuity and visual field development before and after ONSF will be studied. Quality of life assessment will be done before and several times after ONSF.

ELIGIBILITY:
Inclusion Criteria:

* Documented progressive visual function loss over 2 years (visual field or visual acuity)
* Intraocular pressure measured as a maximum of 25 mmHg
* Possibility of receiving general anaesthesia and optic nerve sheath fenestration.

Exclusion Criteria:

* Secondary glaucoma
* Oral medication to lower intraocular pressure (carboanhydrase inhibitor)
* Visual acuity worse than 20/400
* Any other type of glaucoma (pseudoexfoliation, narrow or closed angle).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-03; Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Visual acuity
Visual field
Quality of life assessment
Laboratory markers work-up

CONTACTS AND LOCATIONS:
Overall Officials: Hanspeter E Killer, MD, Prof, Principal Investigator — Kantonsspital Aarau, Department of ophthalmology
Locations (1):
- Kantonsspital Aarau, Department of Ophthalmology, Switzerland, Aarau, Canton of Aargau, Switzerland

REFERENCES:
- [Background] Wax MB, Barrett DA, Hart WM Jr, Custer PL. Optic nerve sheath decompression for glaucomatous optic neuropathy with normal intraocular pressure. Arch Ophthalmol. 1993 Sep;111(9):1219-28. doi: 10.1001/archopht.1993.01090090071022. PMID 8363465
- [Derived] Jaggi GP, Miller NR, Flammer J, Weinreb RN, Remonda L, Killer HE. Optic nerve sheath diameter in normal-tension glaucoma patients. Br J Ophthalmol. 2012 Jan;96(1):53-6. doi: 10.1136/bjo.2010.199224. Epub 2011 Mar 11. PMID 21398413
- See also: Kantonsspital Aarau, Aargau, Switzerland — http://www.ksa.ch